CLINICAL TRIAL: NCT01633489
Title: An Observational Disease and Clinical Outcomes Registry of Patients With Lysosomal Acid Lipase (LAL) Deficiency
Brief Title: Lysosomal Acid Lipase (LAL) Deficiency Registry
Acronym: ALX-LALD-501
Status: Recruiting | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALX-LALD-501
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Lysosomal Acid Lipase Deficiency; Cholesterol Ester Storage Disease; Wolman Disease; Acid Cholesteryl Ester Hydrolase Deficiency, Type 2; Acid Lipase Deficiency; LIPA Deficiency; LAL-Deficiency
MeSH Terms: conditions — Wolman Disease; Cholesterol Ester Storage Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LAL Deficiency patients: Patients are those with a diagnosis of LAL Deficiency (living and deceased), irrespective of treatment status or treatment choice.

SUMMARY:
This is an observational, multi-center, international disease registry designed to collect longitudinal data and create a knowledge base that will be utilized to improve the care and treatment of patients with LAL Deficiency. Participation in the Registry by both physicians and patients is voluntary.

DETAILED DESCRIPTION:
Lysosomal Acid Lipase (LAL) Deficiency is a rare autosomal recessive lysosomal storage disorder (LSD) that is caused by a marked decrease of lysosomal acid lipase (LAL), the enzyme that breaks down cholesteryl esters and triglycerides in the lysosomes.

Lysosomal Acid Lipase Deficiency presenting in infants (historically called Wolman Disease) is a medical emergency with rapid disease progression over a period of weeks that is typically fatal within the first 6 months of life. More commonly, LAL Deficiency presents in children and adults and this presentation has been historically called Cholesteryl Ester Storage Disease (CESD). In general, data on the prevalence of LAL Deficiency are limited, and the overall prevalence of the disease in the population is unclear.

For all presentations, LAL Deficiency is associated with significant morbidity and mortality. Deficient LAL enzyme activity results in the lysosomal accumulation of cholesteryl esters and triglycerides. In the liver, this accumulation leads to hepatomegaly, increased hepatic fat content, transaminase elevation signaling chronic liver injury, and progression to fibrosis, cirrhosis, and complications of end stage liver disease. In the spleen, LAL Deficiency results in splenomegaly, anemia, and thrombocytopenia. Lipid accumulation in the intestinal wall leads to malabsorption and growth failure. Dyslipidemia is common with elevated low density lipoprotein (LDL) and triglycerides and low high density lipoprotein (HDL), associated with increased liver fat content and transaminase elevations. In addition to liver disease, patients with LAL Deficiency experience increased risk for cardiovascular disease and accelerated atherosclerosis.

The LAL Deficiency Registry is a global registry, established to help improve care for patients through improved understanding of the disease and long-term effectiveness of therapeutic interventions including sebelipase alfa.

As with other registries, which are becoming increasingly valuable for collecting information in large, heterogeneous, 'real world' populations, the LAL Deficiency Registry aims to provide evidence to help support patient care and inform clinical practice. This Registry is also being conducted, in part, to fulfill post-marketing commitments and requirements agreed to by the Sponsor as a condition for sebelipase alfa approval in the EU and the USA.

ELIGIBILITY:
Patients must have a confirmed diagnosis of LAL Deficiency. An Informed Consent and Authorization must be obtained prior to patient enrollment where required under applicable laws and regulations, or a waiver must be obtained by the Institutional Review Board/Independent Ethics Committee.

Patients cannot be currently participating in an Alexion-sponsored clinical trial. Patients who have concluded participation in an Alexion-sponsored sebelipase alfa clinical trial are eligible to enroll in this Registry, and enrollment in the Registry will not exclude a patient from enrolling in a future clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a diagnosis of LAL Deficiency.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-05-30 (Actual); Primary Completion 2029-08-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
Understanding of the variability, progression, identification and natural history of LAL Deficiency. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Alexion Pharmaceuticals, Study Director — Sponsor GmbH
Locations (91):
- United States (17):
  - Clinical Trial Site, Phoenix, Arizona
  - Clinical Trial Site, Stanford, California
  - Clinical Trial Site, Miramar, Florida
  - Clinical Trial Site, Orlando, Florida
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Detroit, Michigan
  - Clinical Trial Site, Minneapolis, Minnesota
  - Clinical Trial Site, Jackson, Mississippi
  - Clinical Trial Site, Hackensack, NJ, 7601, New Jersey
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, The Bronx, New York
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, Snyder, Texas
  - Clinical Trial Site, Tacoma, Washington
- Clinical Trial Site, New Lambton Heights, New South Wales, Australia
- Clinical Trial Site, Ghent, East Flanders, Belgium
- Brazil (2):
  - Clinical Trial Site, Campinas, São Paulo
  - Clinical Trial Site, São Paulo
- Clinical Trial Site, Sofia, Sofia-Grad, Bulgaria
- Canada (4):
  - Clinical Trial Site, Edmonton, Alberta
  - Clinical Trial Site, Halifax, Nova Scotia
  - Clinical Trial Site, London, Ontario
  - Clinical Trial Site, Québec
- Clinical Trial Site, Zagreb, Croatia
- Czechia (2):
  - Clinical Trial Site, Prague, Central Bohemia
  - Clinical Trial Site, Olomouc
- France (10):
  - Clinical Trial Site, Bron, Auvergne-Rhône-Alpes
  - Clinical Trial Site, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - Clinical Trial Site, Grenoble, Auvergne-Rhône-Alpes
  - Clinical Trial Site, Caen, Normandy
  - Clinical Trial Site, La Rochelle, Nouvelle-Aquitaine
  - Clinical Trial Site, Niort, Nouvelle-Aquitaine
  - Clinical Trial Site, Nancy, Vandœuvre-lès-Nancy
  - Clinical Trial Site, Dijon
  - Clinical Trial Site, Nantes
  - Clinical Trial Site, Paris, Île-de-France Region
- Germany (4):
  - Clinical Trial Site, Munich, Bavaria
  - Clinical Trial Site, Essen, North Rhine-Westphalia
  - Clinical Trial Site, Mainz, Rhineland-Palatinate
  - Clinical Trial Site, Berlin
- Greece (3):
  - Clinical Trial Site, Athens, Attica
  - Clinical Trial Site, Ioannina, Epirus
  - Clinical Trial Site, Thessaloniki, Macedonia
- Clinical Trial Site, Dublin, Leinster, Ireland
- Israel (3):
  - Clinical Trial Site, Petah Tikva, Central District
  - Clinical Trial Site, Haifa
  - Clinical Trial Site, Jerusalem
- Italy (9):
  - Clinical Trial Site, Bari, Apulia
  - Clinical Trial Site, Napoli, Campania
  - Clinical Trial Site, Udine, Friuli Venezia Giulia
  - Clinical Trial Site, Genoa, Liguria
  - Clinical Trial Site, Bergamo, Lombardy
  - Clinical Trial Site, Milan, Lombardy
  - Clinical Trial Site, Turin, Piedmont
  - Clinical Trial Site, Florence, Tuscany
  - Clinical Trial Site, Padua, Veneto
- Mexico (3):
  - Clinical Trial Site, Zapopan, Jalisco
  - Clinical Trial Site, Aguascalientes
  - Clinical Trial Site, Mexico City
- Clinical Trial Site, Amsterdam, North Holland, Netherlands
- Portugal (2):
  - Clinical Trial Site, Guimarães, Braga District
  - Clinical Trial Site, Lisbon
- Russia (3):
  - Clinical Trial Site, Petersburg, Leningradskaya Oblast'
  - Clinical Trial Site, Moscow, Moscow Oblast
  - Clinical Trial Site, Nizhny Novgorod, Nizhny Novgorod Oblast
- Clinical Trial Site, Riyadh, Saudi Arabia
- Clinical Trial Site, Ljubljana, Slovenia
- Spain (16):
  - Clinical Trial Site, Santiago de Compostela, A Coruña
  - Clinical Trial Site, Barakaldo, Biscay
  - Clinical Trial Site, Logroño, La Rioja
  - Clinical Trial Site, Burela de Cabo, Lugo
  - Clinical Trial Site, Málaga, Málaga
  - Clinical Trial Site, Oviedo, Principality of Asturias
  - Clinical Trial Site, Reus, Tarragona
  - Clinical Trial Site, A Coruña
  - Clinical Trial Site, Albacete
  - Clinical Trial Site, Alicante
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Las Palmas
  - Clinical Trial Site, Madrid
  - Clinical Trial Site, Murcia
  - Clinical Trial Site, Valladolid
  - Clinical Trial Site, Zaragoza
- United Kingdom (5):
  - Clinical Trial Site, Cambridge, Cambridgeshire
  - Clinical Trial Site, London, Greater London
  - Clinical Trial Site, Manchester, Greater Manchester
  - Clinical Trial Site, Salford, Greater Manchester
  - Clinical Trial Site, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Antiga L, Evans J, Ros E, Abel F, Balwani M, Wilson DP, Balistreri W. Sebelipase Alfa Improves Aminotransferase Levels in Lysosomal Acid Lipase Deficiency: Data From an International Registry. Liver Int. 2025 Sep;45(9):e70279. doi: 10.1111/liv.70279. PMID 40781810
- [Derived] Balwani M, Balistreri W, D'Antiga L, Evans J, Ros E, Abel F, Wilson DP. Lysosomal acid lipase deficiency manifestations in children and adults: Baseline data from an international registry. Liver Int. 2023 Jul;43(7):1537-1547. doi: 10.1111/liv.15620. Epub 2023 May 24. PMID 37222260
- [Derived] Soll D, Spira D, Hollstein T, Haberbosch L, Demuth I, Steinhagen-Thiessen E, Bobbert T, Spranger J, Kassner U. Clinical outcome of a patient with lysosomal acid lipase deficiency and first results after initiation of treatment with Sebelipase alfa: A case report. Mol Genet Metab Rep. 2019 Jun 18;20:100479. doi: 10.1016/j.ymgmr.2019.100479. eCollection 2019 Sep. PMID 31249784
- See also: LAL Deficiency Registry — http://www.laldeficiencyregistry.com/
- See also: Alexion Website — http://alexion.com